CLINICAL TRIAL: NCT07038772
Title: Comparison of the Effects of Different Orthodontic Treatment Techniques on Eating Attitudes
Brief Title: Eating Attitudes in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Seda Sağoğlu, Research assistant, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/558
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Eating Behaviors
Keywords: EAT-40; eating attitude; fixed appliance; clear aligner
MeSH Terms: conditions — Feeding Behavior | interventions — Orthodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clear Aligner Treatment (Experimental): Patients undergoing orthodontic treatment with clear aligners
  Interventions: Other: Orthodontic treatment
- Fixed Aligner Treatment (Experimental): Patients undergoing orthodontic treatment with fixed appliance
  Interventions: Other: Orthodontic treatment

INTERVENTIONS:
Other: Orthodontic treatment — Undergoing orthodontic treatment

SUMMARY:
This study was conducted on 70 individuals who presented to the Orthodontics Department of the Faculty of Dentistry at Necmettin Erbakan University. The Eating Attitudes Test (EAT-40) was administered to all patients at the beginning of their treatment (T1) and at the sixth month of treatment (T2), and they were asked to complete it.

DETAILED DESCRIPTION:
This study was conducted on 70 individuals who presented to the Orthodontics Department of the Faculty of Dentistry at Necmettin Erbakan University. Thirty-five patients were randomly selected to receive treatment with clear aligners, while the remaining 35 patients were treated with fixed orthodontic appliances. The Eating Attitudes Test (EAT-40) was administered at the beginning of treatment (T1) and at the sixth month of treatment (T2). Patients were asked to arrive at the clinic half an hour before their appointments to complete the questionnaire. The aim was to evaluate the effect of the type of orthodontic treatment on eating attitudes and behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years,
2. dental Class I, II, or III malocclusion without skeletal discrepancy,
3. absence of impacted or missing teeth,
4. no history of orthodontic treatment,
5. indication for non-extraction orthodontic treatment,
6. Dental Aesthetic Index (DAI) score between 26 and 30,¹⁸
7. no systemic disease or related medication use

Exclusion Criteria:

1. cleft lip/palate,
2. severe temporomandibular joint (TMJ) disorders,
3. poor oral hygiene

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
The change in EAT score over 6 months | 6 months
  If the score is above 30, eating behavior is considered to be negatively affected.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Sağoğlu, Research Assistant, Principal Investigator — Konya Necmettin Erbaka University Faculty of Dentistry
Locations (1):
- Necmettin Erbakan University, Meram, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garner DM, Garfinkel PE. The Eating Attitudes Test: an index of the symptoms of anorexia nervosa. Psychol Med. 1979 May;9(2):273-9. doi: 10.1017/s0033291700030762. PMID 472072
- See also: The Eating Attitudes Test — https://pubmed.ncbi.nlm.nih.gov/?term=The+Eating+Attitudes+Test%3A+an+index+of+the+symptoms+of+anorexia+nervosa
- Available data/document: Study Protocol: EAT-40 — https://www.eat-26.com/